CLINICAL TRIAL: NCT03732066
Title: Web basEd soCial Media tecHnology to Improvement in Adherence to Dual anTiplatelet Therapy Following Drug-Eluting Stent Implantation (WeChat), a Randomized Controlled Branch on Antiplatelet of RESCIND Study
Brief Title: Web basEd soCial Media tecHnology to Improvement in Adherence to Dual anTiplatelet Therapy Following Drug-Eluting Stent Implantation
Acronym: WeChat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Dongguan People's Hospital (Other Government); First People's Hospital, Shunde China (Other); Guangzhou Panyu Central Hospital (Other); Maoming People's Hospital (Other)
Responsible Party: Principal Investigator, Liu yong, Director, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: GDREC2018327H
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Coronary Disease
Keywords: Dual antiplatelet therapy; Mobile health; Discontinuation rate; Drug-eluting stent implantation; Randomized controlled trial
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: Randomization will be performed using a centralized, computerized randomization program in a uniform 1:1 allocation ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients (but not their care providers), research personnel, and investigators will be unaware of their allocation. Study coordinators and research assistants conducting the assessments and statisticians will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive usual text messages, personalized reminders and interactive responses.
  Interventions: Behavioral: Usual Text Messages; Behavioral: Personalized Reminders; Behavioral: Interactive Responses
- Control Group (Other): The control group will receive usual text messages only.
  Interventions: Behavioral: Usual Text Messages

INTERVENTIONS:
Behavioral: Usual Text Messages — Usual text messages four times a week, including cardiovascular knowledge and follow-up reminders, such as risk factors for CHD and typical symptoms of myocardial infarction.
Behavioral: Personalized Reminders — 1. The mHealth tools will provide special interventions according to the patients' medical history. For example, patients with hypertension will receive daily reminders on blood pressure measurement and medication. They will also receive early warning on hypertension with a systolic blood pressure of >180 mmHg or <90 mmHg. Patients who smoke will be required to quit smoking. Every patient will receive a Health Report monthly, which will reflect their drug compliance, blood pressure and so on.
  2. Drug Reminders: Patients' medication information will be recorded by obtaining pictures of their medication. Patients will be asked to punch time clocks simply in the mHealth tools. If they forget to punch cards, they can punch cards whenever they think of it. If there is no record of medication for 3 days, SMS alerts will be received, and phone calls will be received over 7 days.
  Arms: Intervention Group
Behavioral: Interactive Responses — 1. Auto-Response: After sending personal or discomfort symptom questions, the patients will be provided with an automatic response pushed by the back-end database by crawling the keywords. It is suggested that the answer is just for reference. In case of urgent questions, they will be advised to consult the clinicians.
  2. The researchers will communicate with the patients every month.
  Arms: Intervention Group

SUMMARY:
Few studies have attempt to improve DAPT adherence through social media. The investigators will explore the prevalence of DAPT discontinuation and prove the hypothesis that using social media will improve DAPT adherence among patients requiring DAPT following DES implantation.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) is frequently discontinued after drug-eluting stent (DES) implantation, which could lead to many major adverse cardiovascular events (MACEs). Social media have been proven effective in improving lifestyles and blood pressures control, but few studies have attempt to improve DAPT adherence through social media.Therefore, eligible patients will be enrolled through scanning QR code and randomized in a 1:1 ratio to an intervention group or control group with 12 months of follow-up.The investigators will find out the prevalence of DAPT discontinuation and prove the hypothesis that using social media will improve DAPT adherence among patients requiring DAPT following DES implantation..

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* diagnosed CHD and underwent DES implantation
* provide written informed consent

Exclusion Criteria:

* pregnancy
* malignant tumor or end-stage disease with a life expectancy of <1 year;
* refusal to use social media
* refusal to provide written informed consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Discontinuation of Dual Antiplatelet Drug | 1 year
  Defined as discontinuation of any dual antiplatelet drug owing to patients' own discretion, including bleeding or non-compliance rather than doctors' advice. Changing of DAPT medication between ticagrelor and clopidogrel under doctors' advice will not be identified as dual antiplatelet drug discontinuation; changing of such under own discretion will be identified as such

SECONDARY OUTCOMES:
Medication Adherence | 1 year
  Dual antiplatelet therapy (DAPT) adherence according to proportion of days covered (PDC) by prescription.
Number of Participants with Major Adverse Cardiovascular Events | 1 year
  All-cause mortality,target vessel revascularization, non-fatal myocardial infarction, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD, Study Chair — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Sun GL, Lei L, Liu L, Liu J, He Y, Guo Z, Dai X, He L, Chen SQ, Liang Y, Ye J, Hu Y, Chen G, Chen JY, Liu Y. Rationale and design of the Web-basEd soCial media tecHnology to improvement in Adherence to dual anTiplatelet Therapy following Drug-Eluting Stent Implantation (WECHAT): protocol for a randomised controlled study. BMJ Open. 2020 Jan 7;10(1):e033017. doi: 10.1136/bmjopen-2019-033017. PMID 31915170